CLINICAL TRIAL: NCT04225715
Title: A Phase II, Randomised, Adaptive, Open-Label Platform Trial To Evaluate Efficacy And Safety Of Multiple Combination Therapies In Participants With Chronic Hepatitis B
Brief Title: A Trial To Evaluate The Efficacy And Safety Of Multiple Combination Therapies In Participants With Chronic Hepatitis B
Acronym: Piranga
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WV41073; 2019-002086-35 (EudraCT Number)
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Results first posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — linvencorvir; RO7020531; RNA, Small Interfering; peginterferon alfa-2a

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Nucleos(t)ide (NUC) Control Arm (Active Comparator): Participants will continue their background NUC therapy for the 48-week treatment period. At the end of the treatment period, in line with current CHB treatment guidelines, participants will continue NUC treatment during the follow-up unless the NUC discontinuation criteria have been met.
  Interventions: Drug: Nucleos(t)ide (NUC)
- Core Protein Allosteric Modulator (CpAM; RO7049389) + Toll-like Receptor 7 (TLR7;RO7020531) + NUC (Experimental): Participants will receive RO7049389 (600 mg once daily [QD]) in addition to their background NUC therapy for the 48-week treatment period. RO7020531 (150 mg once every other day [QOD]) will be administered during Weeks 1-12 and Weeks 25-36. At the end of the treatment period, participants will continue NUC treatment during the follow-up unless the NUC discontinuation criteria have been met.
  Interventions: Drug: Nucleos(t)ide (NUC); Drug: CpAM (RO7049389); Drug: TLR7 (RO7020531)
- Short Interfering Ribonucleic acid (siRNA; RO7445482) (Dose1) + NUC (Experimental): Participants will receive RO7445482 (Dose 1) in addition to their background NUC therapy for the 48-week treatment period. At the end of the treatment period, participants will continue NUC treatment during the follow-up unless the NUC discontinuation criteria have been met.
  Interventions: Drug: Nucleos(t)ide (NUC); Drug: siRNA (RO7445482)
- siRNA (RO7445482) (Dose 2) + NUC (Experimental): Participants will receive RO7445482 (Dose 2) in addition to their background NUC therapy for the 48-week treatment period. At the end of the treatment period, participants will continue NUC treatment during the follow-up unless the NUC discontinuation criteria have been met.
  Interventions: Drug: Nucleos(t)ide (NUC); Drug: siRNA (RO7445482)
- siRNA (RO7445482) + Pegylated Interferon (PEG-IFN) + NUC (Experimental): Participants will receive RO7445482 (Dose 2) in addition to their background NUC therapy for the 48-week treatment period. PEG-IFN will be administered at a dose of 180 μg once weekly (QW) for 48 weeks. At the end of the treatment period, participants will continue NUC treatment during the follow-up unless the NUC discontinuation criteria have been met.
  Interventions: Drug: Nucleos(t)ide (NUC); Drug: siRNA (RO7445482); Drug: PEG-IFN
- siRNA (RO7445482) + CpAM (RO7049389) + NUC (Experimental): Participants will receive RO7445482 (Dose 2) and RO7049389 (600 mg QD) in addition to their background NUC therapy for the 48-week treatment period. At the end of the treatment period, participants will continue NUC treatment during the follow-up unless the NUC discontinuation criteria have been met.
  Interventions: Drug: Nucleos(t)ide (NUC); Drug: CpAM (RO7049389); Drug: siRNA (RO7445482)
- siRNA (RO7445482) + TLR7 (RO7020531) + NUC (Experimental): Participants will receive RO7445482 (Dose 2) in addition to their background NUC therapy for the 48-week treatment period. RO7020531 (150 mg QOD) will be administered during Weeks 13-24 and Weeks 37-48 (i.e., 2 treatment cycles of 12 weeks' duration each and 42 doses of RO7020531 for each cycle). At the end of the treatment period, participants will continue NUC treatment during the follow-up unless the NUC discontinuation criteria have been met.
  Interventions: Drug: Nucleos(t)ide (NUC); Drug: TLR7 (RO7020531); Drug: siRNA (RO7445482)
- siRNA(RO7445482)+ Programmed Death Ligand-1 Locked Nucleic Acid (PD-L1 LNA; RO7191863) + NUC [1] (Experimental): Participants will receive RO7445482 (Dose 2) during Weeks 1-24 and RO7191863 (Dose 1) will be administered during Weeks 13-24, in addition to their background NUC therapy for the 24-week treatment period. At the end of the treatment period, participants will continue NUC treatment during the follow-up unless the NUC discontinuation criteria have been met.
  Interventions: Drug: Nucleos(t)ide (NUC); Drug: siRNA (RO7445482); Drug: PD-L1 LNA (RO7191863)
- siRNA (RO7445482) + PD-L1 LNA (RO7191863) + NUC [2] (Experimental): Participants will receive RO7445482 (Dose 2) during Weeks 1-24 and RO7191863 (Dose 1) will be administered during Weeks 25-36, in addition to their background NUC therapy for the 36-week treatment period. At the end of the treatment period, participants will continue NUC treatment during the follow-up unless the NUC discontinuation criteria have been met.
  Interventions: Drug: Nucleos(t)ide (NUC); Drug: siRNA (RO7445482); Drug: PD-L1 LNA (RO7191863)

INTERVENTIONS:
Drug: Nucleos(t)ide (NUC) — Nucleos(t)ide (NUC) will be administered orally
Drug: CpAM (RO7049389) — CpAM (RO7049389) will be administered orally
  Other Names: Linvencorvir; RG7907
  Arms: Core Protein Allosteric Modulator (CpAM; RO7049389) + Toll-like Receptor 7 (TLR7;RO7020531) + NUC; siRNA (RO7445482) + CpAM (RO7049389) + NUC
Drug: TLR7 (RO7020531) — TLR7 (RO7020531) will be administered orally
  Other Names: Ruzotolimod; RG7854
  Arms: Core Protein Allosteric Modulator (CpAM; RO7049389) + Toll-like Receptor 7 (TLR7;RO7020531) + NUC; siRNA (RO7445482) + TLR7 (RO7020531) + NUC
Drug: siRNA (RO7445482) — siRNA (RO7445482) will be administered subcutaneously
  Other Names: Xalnesiran; RG6346
  Arms: Short Interfering Ribonucleic acid (siRNA; RO7445482) (Dose1) + NUC; siRNA (RO7445482) (Dose 2) + NUC; siRNA (RO7445482) + CpAM (RO7049389) + NUC; siRNA (RO7445482) + PD-L1 LNA (RO7191863) + NUC [2]; siRNA (RO7445482) + Pegylated Interferon (PEG-IFN) + NUC; siRNA (RO7445482) + TLR7 (RO7020531) + NUC; siRNA(RO7445482)+ Programmed Death Ligand-1 Locked Nucleic Acid (PD-L1 LNA; RO7191863) + NUC [1]
Drug: PEG-IFN — PEG-IFN will be administered subcutaneously
  Other Names: Pegasys®
  Arms: siRNA (RO7445482) + Pegylated Interferon (PEG-IFN) + NUC
Drug: PD-L1 LNA (RO7191863) — PD-L1 LNA (RO7191863) will be administered subcutaneously
  Other Names: Cadapersen; RG6084
  Arms: siRNA (RO7445482) + PD-L1 LNA (RO7191863) + NUC [2]; siRNA(RO7445482)+ Programmed Death Ligand-1 Locked Nucleic Acid (PD-L1 LNA; RO7191863) + NUC [1]

SUMMARY:
This is a study designed to evaluate the safety, tolerability and efficacy of New Molecular Entity (NME) combination therapies in Chronic Hepatitis B (CHB) participants with preserved liver function and without significant fibrosis/cirrhosis. The platform design allows comparison of multiple NME combination therapies against a common control, and introduction of additional treatment arms at later study time points. Each arm will consist of a screening phase (up to 8 weeks), treatment phase (up to 48 weeks) and post-treatment follow-up phase (48 weeks). The safety and efficacy will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18 and 32 kg/m2 inclusive.
* Participants with Chronic Hepatitis B (CHB) infection (HBsAg positive for >=6 months) who are on established NUC (entecavir or tenofovir alafenamide/disoproxil fumarate) monotherapy for >=12 months, having received the same NUC therapy for >=3 months prior to screening.
* HBV DNA below the lower LLOQ or < 20 IU/mL for > 6 months prior to screening and confirmed at screening.
* Alanine transaminase (ALT) <=1.5 x upper limit of normal (ULN) for > 6 months prior to screening and confirmed at screening.
* Female Participants: Eligible to participate if she is not pregnant, not breastfeeding and agrees to remain abstinent (refrain from heterosexual intercourse) or use highly effective contraceptive methods.
* Male Participants: During the treatment period and for at least 6 months after the final dose of study treatment, agrees to remain abstinent (refrain from heterosexual intercourse), use contraceptive measures and refrain from donating sperm.

Exclusion Criteria:

* Pregnant or lactating women.
* Co-infection with other pathogens such as Hepatitis A, C, D and E or Human Immunodeficiency Virus (HIV).
* History of cirrhosis or current evidence of significant liver fibrosis or cirrhosis or decompensated liver disease.
* History of or suspicion of Hepatocellular Carcinoma (HCC).
* Thyroid disease poorly controlled on prescribed medications or clinically relevant abnormal thyroid function tests.
* Clinically significant disease other than CHB that, in the opinion of the Investigator, makes the participant unsuitable for the study.
* Pre-existing cardiac disease that in the opinion of the investigator would increase the risk for the participant to take part in the study.
* History of alcohol abuse and/or drug abuse within one year of randomization.
* History of having received (in the last 6 months) or currently receiving any systemic antineoplastic (including radiation) or immunosuppressive (including biologic immunosuppressors) or immune modulating treatment.
* Currently taking, or have received within 3 months of Day 1, systemic corticosteroids.
* Electrocardiogram (ECG) with clinically significant abnormalities.
* Previous treatment with an investigational agent for Hepatitis B (HBV) within 6 months prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2020-07-05 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (33):
- Bulgaria (2):
  - Tokuda Hospital Sofia, Sofia
  - University Multiprofile Hospital For Active Treatment "Sveti Ivan Rilski" EAD, Sofia
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - Uni of Alberta Hospital, Edmonton, Alberta
  - Toronto Liver Centre, Toronto, Ontario
- Hospital San Juan de Dios La Serena, La Serena, Chile
- China (6):
  - Beijing Friendship Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Huashan Hospital, Fudan University, Shanghai
- Hopital Beaujon, Clichy, France
- Queen Mary Hospital, Hong Kong, Hong Kong
- New Zealand (2):
  - Auckland Clinical Studies Limited, Auckland
  - Middlemore Clinical Trials, Auckland
- Spitalul Clinic Judetean de Urgenta Cluj Napoca, Cluj-Napoca, Romania
- South Korea (4):
  - Chuncheon Sacred Heart Hospital, Gangwon-Do
  - Asan Medical Center / Clinical Trial Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Seoul National University College of Medicine, Liver Research Institute, Seoul
- Spain (2):
  - Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
- Taiwan (6):
  - Changhua Christian Hospital, Chang-hua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung Univ Hosp, Tainan
  - National Taiwan University Hospital, Taipei
- Thailand (3):
  - HIVNAT, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
- King College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Hou J, Zhang W, Xie Q, Hua R, Tang H, Morano Amado LE, Yang SS, Peng CY, Su WW, Chuang WL, Kim DJ, Avihingsanon A, Kao JH, Leerapun A, Yuen MF, Asselah T, Liang X, Bo Q, Canducci F, Catanese MT, Chen E, Cheng C, Chughlay F, Das S, Glavini K, Guerreiro N, Huang Y, Kakrana P, Kazma R, Patil A, Pavlovic V, Surujbally B, Triyatni M, Upmanyu R, Wat C, Gane E; Piranga Study Group. Xalnesiran with or without an Immunomodulator in Chronic Hepatitis B. N Engl J Med. 2024 Dec 5;391(22):2098-2109. doi: 10.1056/NEJMoa2405485. PMID 39774313

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 281 participants with chronic hepatitis B (CHB) who had virologic suppression with Nucleos(t)ide (NUC) therapy took part in the study across 13 countries from 05 July 2020 to 19 July 2024.
Pre-assignment Details: The study consisted of a screening phase, followed by up to 48 weeks of treatment and up to 48 weeks of post-treatment follow-up. Multiple new combination therapies were compared against a common control. Combos 1, 5, 7 and 8 were prematurely terminated by the Sponsor.
Groups:
- NUC Control Arm: Participants continued their background NUC therapy for 48 weeks. Thereafter, in line with current CHB treatment guidelines, participants continued NUC treatment during follow-up unless the NUC discontinuation criteria were met.
- Combo 1: CpAM + TLR7 Agonist + NUC: Participants received core protein allosteric modulator (CpAM), 600 milligrams (mg) tablets, orally, once daily (QD) for 48 weeks and toll-like receptor 7 (TLR7) agonist, 150 mg, orally, once every other day (QOD) during Weeks 1-12 and Weeks 25-36 in addition to their background NUC therapy. After Week 48, participants continued NUC treatment during follow-up unless the NUC discontinuation criteria were met.
- Combo 2: siRNA (100 mg) + NUC: Participants received short interfering ribonucleic acid (siRNA), 100 mg, as a subcutaneous (SC) injection, every 4 weeks (Q4W) in addition to their background NUC therapy for 48 weeks. After Week 48, participants continued NUC treatment during follow-up unless the NUC discontinuation criteria were met.
- Combo 3: siRNA (200 mg) + NUC: Participants received siRNA, 200 mg, as a SC injection, Q4W in addition to their background NUC therapy for 48 weeks. After Week 48, participants continued NUC treatment during follow-up unless the NUC discontinuation criteria were met.
- Combo 4: siRNA + PEG-IFN + NUC: Participants received siRNA, 200 mg, as a SC injection, Q4W and pegylated interferon (PEG-IFN), 180 micrograms (µg), as a SC injection, every week (QW) in addition to their background NUC therapy for 48 weeks. After Week 48, participants continued NUC treatment during follow-up unless the NUC discontinuation criteria were met.
- Combo 5: siRNA + CpAM + NUC: Participants received siRNA, 200 mg, as a SC injection, Q4W and CpAM, 600 mg tablets, orally, QD in addition to their background NUC therapy for 48 weeks. After Week 48, participants continued NUC treatment during follow-up unless the NUC discontinuation criteria were met.
- Combo 6: siRNA + TLR7 Agonist + NUC: Participants received siRNA, 200 mg, as a SC injection, Q4W for 48 weeks and TLR7 agonist, 150 mg tablets, orally, QOD during Weeks 13-24 and Weeks 37-48 in addition to their background NUC therapy. After Week 48, participants continued NUC treatment during follow-up unless the NUC discontinuation criteria were met.
- Combo 7: siRNA + PD-L1 LNA + NUC: Participants received siRNA, 200 mg, as a SC injection, Q4W up to Week 24 and programmed death ligand-1 locked nucleic acid (PD-L1 LNA), 2 milligrams/kilograms (mg/kg), as a SC injection, QW during Weeks 13-24 in addition to their background NUC therapy for 24 weeks. After Week 24, participants continued NUC treatment during follow-up unless the NUC discontinuation criteria were met.
- Combo 8: siRNA + PD-L1 LNA + NUC: Participants received siRNA, 200 mg, as a SC injection, Q4W up to Week 24 and PD-L1 LNA, 2 mg/kg, as a SC injection, QW during Weeks 25-36 in addition to their background NUC therapy for 36 weeks. After Week 36, participants continued NUC treatment during follow-up unless the NUC discontinuation criteria were met.
Period: Overall Study
Arm/Group | NUC Control Arm | Combo 1: CpAM + TLR7 Agonist + NUC | Combo 2: siRNA (100 mg) + NUC | Combo 3: siRNA (200 mg) + NUC | Combo 4: siRNA + PEG-IFN + NUC | Combo 5: siRNA + CpAM + NUC | Combo 6: siRNA + TLR7 Agonist + NUC | Combo 7: siRNA + PD-L1 LNA + NUC | Combo 8: siRNA + PD-L1 LNA + NUC
Started | 36 | 38 | 30 | 30 | 30 | 19 | 34 | 33 | 31
Completed | 30 | 37 | 29 | 30 | 27 | 9 | 33 | 15 | 12
Not Completed | 6 | 1 | 1 | 0 | 3 | 10 | 1 | 18 | 19
Not completed — Reason not Specified | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 9 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 1 | 0 | 3 | 1 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Arm Terminated By Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 18

BASELINE CHARACTERISTICS:
Population: All participants population included all participants who were randomized to their treatment regimen.
Groups:
- Combo 1: CpAM + TLR7 Agonist + NUC: Participants received CpAM, 600 mg tablets, orally, QD for 48 weeks and TLR7 agonist, 150 mg, orally, QOD during Weeks 1-12 and Weeks 25-36 in addition to their background NUC therapy. After Week 48, participants continued NUC treatment during follow-up unless the NUC discontinuation criteria were met.
- Combo 2: siRNA (100 mg) + NUC: Participants received siRNA, 100 mg, as a SC injection, Q4W in addition to their background NUC therapy for 48 weeks. After Week 48, participants continued NUC treatment during follow-up unless the NUC discontinuation criteria were met.
- Combo 4: siRNA + PEG-IFN + NUC: Participants received siRNA, 200 mg, as a SC injection, Q4W and PEG-IFN, 180 µg, as a SC injection, QW in addition to their background NUC therapy for 48 weeks. After Week 48, participants continued NUC treatment during follow-up unless the NUC discontinuation criteria were met.
- Combo 7: siRNA + PD-L1 LNA + NUC: Participants received siRNA, 200 mg, as a SC injection, Q4W up to Week 24 and PD-L1 LNA, 2 mg/kg, as a SC injection, QW during Weeks 13-24 in addition to their background NUC therapy for 24 weeks. After Week 24, participants continued NUC treatment during follow-up unless the NUC discontinuation criteria were met.
- Total: Total of all reporting groups
Arm/Group | NUC Control Arm | Combo 1: CpAM + TLR7 Agonist + NUC | Combo 2: siRNA (100 mg) + NUC | Combo 3: siRNA (200 mg) + NUC | Combo 4: siRNA + PEG-IFN + NUC | Combo 5: siRNA + CpAM + NUC | Combo 6: siRNA + TLR7 Agonist + NUC | Combo 7: siRNA + PD-L1 LNA + NUC | Combo 8: siRNA + PD-L1 LNA + NUC | Total
Number analyzed (Participants) | 36 | 38 | 30 | 30 | 30 | 19 | 34 | 33 | 31 | 281
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 36 | 38 | 28 | 29 | 30 | 19 | 34 | 33 | 30 | 277
  >=65 years | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 1 | 10 | 5 | 5 | 4 | 10 | 6 | 58
  Male | 28 | 29 | 29 | 20 | 25 | 14 | 30 | 23 | 25 | 223
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 35 | 37 | 30 | 30 | 30 | 19 | 34 | 33 | 30 | 278
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 33 | 34 | 26 | 29 | 30 | 19 | 32 | 22 | 22 | 247
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 5
  White | 2 | 3 | 3 | 1 | 0 | 0 | 0 | 9 | 8 | 26
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hepatitis B Surface Antigen (HBsAg) Loss at 24 Weeks Post-End of Treatment (EOT)
Description: HBsAg loss was defined as quantitative HBsAg <0.05 international units/milliliters (IU/mL). The percentage of participants with HBsAg loss was calculated as number of participants with HBsAg loss / total number of participants *100. 95% confidence interval (CI) was calculated using the Clopper-Pearson method. Percentages have been rounded off.
Time Frame: Follow-up Week (FUW) 24
Population: Modified Intent to Treat (mITT) population included participants who were randomized and received at least one dose of each drug for their assigned treatment regimen. Overall number analyzed included participants with data available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- NUC Control Arm: Participants continued their background NUC therapy for 48 weeks. Thereafter, in line with current CHB treatment guidelines, participants continued NUC treatment during the follow-up unless the NUC discontinuation criteria were met.
- Combo 2: siRNA (100 mg) + NUC: Participants received siRNA, 100 mg, as a SC injection, Q4W in addition to their background NUC therapy for 48 weeks. After Week 48, participants continued NUC treatment during the follow-up unless the NUC discontinuation criteria were met.
- Combo 3: siRNA (200 mg) + NUC: Participants received siRNA, 200 mg, as a SC injection, Q4W in addition to their background NUC therapy for 48 weeks. After Week 48, participants continued NUC treatment during the follow-up unless the NUC discontinuation criteria were met.
- Combo 4: siRNA + PEG-IFN + NUC: Participants received siRNA, 200 mg, as a SC injection, Q4W and PEG-IFN, 180 µg, as a SC injection, QW in addition to their background NUC therapy for 48 weeks. After Week 48, participants continued NUC treatment during the follow-up unless the NUC discontinuation criteria were met.
- Combo 5: siRNA + CpAM + NUC: Participants received siRNA, 200 mg, as a SC injection, Q4W and CpAM, 600 mg tablets, orally, QD in addition to their background NUC therapy for 48 weeks. After Week 48, participants continued NUC treatment during the follow-up unless the NUC discontinuation criteria were met.
- Combo 6: siRNA + TLR7 Agonist + NUC: Participants received siRNA, 200 mg, as a SC injection, Q4W for 48 weeks and TLR7 agonist, 150 mg tablets, orally, QOD during Weeks 13-24 and Weeks 37-48 in addition to their background NUC therapy. After Week 48, participants continued NUC treatment during the follow-up unless the NUC discontinuation criteria were met.
- Combo 7: siRNA + PD-L1 LNA + NUC: Participants received siRNA, 200 mg, as a SC injection, Q4W up to Week 24 and PD-L1 LNA, 2 mg/kg, as a SC injection, QW during Weeks 13-24 in addition to their background NUC therapy for 24 weeks. After Week 24, participants continued NUC treatment during the follow-up unless the NUC discontinuation criteria were met.
- Combo 8: siRNA + PD-L1 LNA + NUC: Participants received siRNA, 200 mg, as a SC injection, Q4W up to Week 24 and PD-L1 LNA, 2 mg/kg, as a SC injection, QW during Weeks 25-36 in addition to their background NUC therapy for 36 weeks. After Week 36, participants continued NUC treatment during the follow-up unless the NUC discontinuation criteria were met.
Arm/Group | NUC Control Arm | Combo 1: CpAM + TLR7 Agonist + NUC | Combo 2: siRNA (100 mg) + NUC | Combo 3: siRNA (200 mg) + NUC | Combo 4: siRNA + PEG-IFN + NUC | Combo 5: siRNA + CpAM + NUC | Combo 6: siRNA + TLR7 Agonist + NUC | Combo 7: siRNA + PD-L1 LNA + NUC | Combo 8: siRNA + PD-L1 LNA + NUC
Number analyzed (Participants) | 35 | 35 | 30 | 30 | 30 | 9 | 34 | 33 | 30
percentage of participants | 0 [0 to 10] | 0 [0 to 0] | 6.7 [0.8 to 22.1] | 3.3 [0.1 to 17.2] | 23.3 [9.9 to 42.3] | 0 [0 to 0] | 11.8 [3.3 to 27.5] | 0 [0 to 10.6] | 6.7 [0.8 to 22.1]
Statistical Analysis 1: Comparison: NUC Control Arm vs Combo 2: siRNA (100 mg) + NUC; Test type: Superiority; Difference in Response Rate = 7.2, 95% CI 2-sided [-2.1 to 16.4] — 95% CI for difference of two proportions was calculated using Cochran-Mantel-Haenszel (CMH) method
Statistical Analysis 2: Comparison: NUC Control Arm vs Combo 3: siRNA (200 mg) + NUC; Test type: Superiority; Difference in Response Rate = 3.5, 95% CI 2-sided [-3.1 to 10] — 95% CI for difference of two proportions was calculated using CMH method
Statistical Analysis 3: Comparison: NUC Control Arm vs Combo 4: siRNA + PEG-IFN + NUC; Test type: Superiority; Difference in Response Rate = 24.3, 95% CI 2-sided [9 to 39.5] — 95% CI for difference of two proportions was calculated using CMH method
Statistical Analysis 4: Comparison: NUC Control Arm vs Combo 6: siRNA + TLR7 Agonist + NUC; Test type: Superiority; Difference in Response Rate = 12.3, 95% CI 2-sided [1.3 to 23.3] — 95% CI for difference of two proportions was calculated using CMH method
Statistical Analysis 5: Comparison: NUC Control Arm vs Combo 7: siRNA + PD-L1 LNA + NUC; Test type: Superiority; Difference in Response Rate = 0, 95% CI 2-sided [0 to 0] — 95% CI for difference of two proportions was calculated using CMH method
Statistical Analysis 6: Comparison: NUC Control Arm vs Combo 8: siRNA + PD-L1 LNA + NUC; Test type: Superiority; Difference in Response Rate = 6.7, 95% CI 2-sided [-2.2 to 15.7] — 95% CI for difference of two proportions was calculated using CMH method

2. Secondary Outcome: Percentage of Participants With HBsAg Loss
Description: HBsAg loss was defined as quantitative HBsAg <0.05 IU/mL. The percentage of participants with HBsAg loss was calculated as number of participants with HBsAg loss / total number of participants *100. 95% CI was calculated using the Clopper-Pearson method. Percentages have been rounded off.
Time Frame: Combos 1 and 5: Weeks 24, 36, 48 and FUW 48; Combos 2, 3, 4, 6 and NUC Arm: Week 48 and FUW 48; Combo 7: Week 24; Combo 8: Week 36
Population: mITT population included participants who were randomized and received at least one dose of each drug for their assigned treatment regimen. Overall number analyzed included participants with data available for analysis. Number analyzed included participants with data available for analysis at that specified timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NUC Control Arm | Combo 1: CpAM + TLR7 Agonist + NUC | Combo 2: siRNA (100 mg) + NUC | Combo 3: siRNA (200 mg) + NUC | Combo 4: siRNA + PEG-IFN + NUC | Combo 5: siRNA + CpAM + NUC | Combo 6: siRNA + TLR7 Agonist + NUC | Combo 7: siRNA + PD-L1 LNA + NUC | Combo 8: siRNA + PD-L1 LNA + NUC
Number analyzed (Participants) | 35 | 36 | 30 | 30 | 30 | 4 | 34 | 33 | 30
percentage of participants
  Week 24: number analyzed (Participants) | 0 | 36 | 0 | 0 | 0 | 4 | 0 | 33 | 0
  Week 24 |  | 0 [0 to 0] |  |  |  | 0 [0 to 0] |  | 6.1 [0.7 to 20.2] |
  Week 36: number analyzed (Participants) | 0 | 23 | 0 | 0 | 0 | 1 | 0 | 0 | 30
  Week 36 |  | 0 [0 to 0] |  |  |  | 0 [0 to 0] |  |  | 13.3 [3.8 to 30.7]
  Week 48: number analyzed (Participants) | 35 | 20 | 30 | 30 | 30 | 4 | 34 | 0 | 0
  Week 48 | 0 [0 to 10] | 0 [0 to 0] | 6.7 [0.8 to 22.1] | 3.3 [0.1 to 17.2] | 30 [14.7 to 49.4] | 0 [0 to 0] | 17.6 [6.8 to 34.5] |  |
  FUW 48: number analyzed (Participants) | 35 | 28 | 30 | 30 | 30 | 1 | 34 | 0 | 0
  FUW 48 | 2.9 [0.1 to 14.9] | 0 [0 to 0] | 10 [2.1 to 26.5] | 0 [0 to 11.6] | 16.7 [5.6 to 34.7] | 0 [0 to 0] | 11.8 [3.3 to 27.5] |  |
Statistical Analysis 1: Comparison: NUC Control Arm vs Combo 7: siRNA + PD-L1 LNA + NUC; Combo 7: Week 24; Test type: Superiority; 6.2 = 6.2, 95% CI 2-sided [-2 to 14.5] — 95% CI for difference of two proportions was calculated using CMH method
Statistical Analysis 2: Comparison: NUC Control Arm vs Combo 8: siRNA + PD-L1 LNA + NUC; Combo 8: Week 36; Test type: Superiority; Difference in Response Rate = 13.4, 95% CI 2-sided [1.2 to 25.6] — 95% CI for difference of two proportions was calculated using CMH method
Statistical Analysis 3: Comparison: NUC Control Arm vs Combo 2: siRNA (100 mg) + NUC; Combo 2: Week 48; Test type: Superiority; Difference in Response Rate = 7.2, 95% CI 2-sided [-2.1 to 16.4] — 95% CI for difference of two proportions was calculated using CMH method
Statistical Analysis 4: Comparison: NUC Control Arm vs Combo 3: siRNA (200 mg) + NUC; Combo 3: Week 48; Test type: Superiority; Difference in Response Rate = 3.5, 95% CI 2-sided [-3.1 to 10] — 95% CI for difference of two proportions was calculated using CMH method
Statistical Analysis 5: Comparison: NUC Control Arm vs Combo 4: siRNA + PEG-IFN + NUC; Combo 4: Week 48; Test type: Superiority; Difference in Response Rate = 31.2, 95% CI 2-sided [14.7 to 47.6] — 95% CI for difference of two proportions was calculated using CMH method
Statistical Analysis 6: Comparison: NUC Control Arm vs Combo 6: siRNA + TLR7 Agonist + NUC; Combo 6: Week 48; Test type: Superiority; Difference in Response Rate = 18.4, 95% CI 2-sided [5.4 to 31.4] — 95% CI for difference of two proportions was calculated using CMH method
Statistical Analysis 7: Comparison: NUC Control Arm vs Combo 2: siRNA (100 mg) + NUC; Combo 2: FUW 48; Test type: Superiority; Difference in Response Rate = 8.1, 95% CI 2-sided [-3.9 to 20.1] — 95% CI for difference of two proportions was calculated using CMH method
Statistical Analysis 8: Comparison: NUC Control Arm vs Combo 3: siRNA (200 mg) + NUC; Combo 3: FUW 48; Test type: Superiority; Difference in Response Rate = -2.7, 95% CI 2-sided [-8.1 to 2.7] — 95% CI for difference of two proportions was calculated using CMH method
Statistical Analysis 9: Comparison: NUC Control Arm vs Combo 4: siRNA + PEG-IFN + NUC; Combo 4: FUW 48; Test type: Superiority; Difference in Response Rate = 14.6, 95% CI 2-sided [0.4 to 28.8] — 95% CI for difference of two proportions was calculated using CMH method
Statistical Analysis 10: Comparison: NUC Control Arm vs Combo 6: siRNA + TLR7 Agonist + NUC; Combo 6: FUW 48; Test type: Superiority; Difference in Response Rate = 9.5, 95% CI 2-sided [-2.5 to 21.5] — 95% CI for difference of two proportions was calculated using CMH method

3. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion
Description: HBsAg seroconversion was defined as a quantitative HBsAg < 0.05 IU/mL and a positive anti-HBs antibody (defined as per assay reactive threshold anti-HBs ≥10 IU/L). 95% CI was calculated using the Clopper-Pearson method. Percentages have been rounded off.
Time Frame: Combos 1 and 5: Weeks 24, 36, 48, FUW 24 and FUW 48; Combos 2, 3, 4, 6 and NUC Arm: Week 48, FUW 24 and FUW 48; Combo 7: Week 24 and FUW 24; Combo 8: Week 36 and FUW 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NUC Control Arm | Combo 1: CpAM + TLR7 Agonist + NUC | Combo 2: siRNA (100 mg) + NUC | Combo 3: siRNA (200 mg) + NUC | Combo 4: siRNA + PEG-IFN + NUC | Combo 5: siRNA + CpAM + NUC | Combo 6: siRNA + TLR7 Agonist + NUC | Combo 7: siRNA + PD-L1 LNA + NUC | Combo 8: siRNA + PD-L1 LNA + NUC
Number analyzed (Participants) | 35 | 36 | 30 | 30 | 30 | 9 | 34 | 33 | 30
percentage of participants
  Week 24: number analyzed (Participants) | 0 | 36 | 0 | 0 | 0 | 9 | 0 | 33 | 0
  Week 24 |  | 0 [0 to 0] |  |  |  | 0 [0 to 0] |  | 0 [0 to 10.6] |
  Week 36: number analyzed (Participants) | 0 | 23 | 0 | 0 | 0 | 1 | 0 | 0 | 30
  Week 36 |  | 0 [0 to 0] |  |  |  | 0 [0 to 0] |  |  | 0 [0 to 11.9]
  Week 48: number analyzed (Participants) | 35 | 20 | 30 | 30 | 30 | 4 | 34 | 0 | 0
  Week 48 | 0 [0 to 10] | 0 [0 to 0] | 3.3 [0.1 to 17.2] | 0 [0 to 11.6] | 23.3 [9.9 to 42.3] | 0 [0 to 0] | 0 [0 to 10.3] |  |
  FUW 24: number analyzed (Participants) | 35 | 35 | 30 | 30 | 30 | 9 | 34 | 33 | 30
  FUW 24 | 0 [0 to 10] | 0 [0 to 0] | 3.3 [0.1 to 17.2] | 0 [0 to 11.6] | 20 [7.7 to 38.6] | 0 [0 to 0] | 3.1 [0.1 to 16.2] | 0 [0 to 10.9] | 0 [0 to 11.6]
  FUW 48: number analyzed (Participants) | 35 | 28 | 30 | 30 | 30 | 1 | 34 | 0 | 0
  FUW 48 | 2.9 [0.1 to 14.9] | 0 [0 to 0] | 3.3 [0.1 to 17.2] | 0 [0 to 11.6] | 16.7 [5.6 to 34.7] | 0 [0 to 0] | 5.9 [0.7 to 19.7] |  |

4. Secondary Outcome: Percentage of Participants With Hepatitis B Early Antigen (HBeAg) Loss in Baseline HBeAg-positive Participants
Description: HBeAg loss was defined as negative /non-reactive HBeAg level. Percentages have been rounded off.
Time Frame: Weeks 12, 24, 36, and 48; FUW 12, 24, 36, and 48
Population: mITT population included participants who were randomized and received at least one dose of each drug for their assigned treatment regimen. Overall number analyzed included participants from the mITT population who were positive for HBeAg at baseline. Number analyzed included participants with data available for analysis at that specified timepoint.
Measure: Number; unit: percentage of participants
Groups:
- Combo 7: siRNA + PD-L1 LNA + NUC: Participants received siRNA, 200 mg, as a SC injection, Q4W up to Week 24 and PD-L1 LNA, 2 mg/kg, as a SC injection, QW during Weeks 13-24 in addition to their background NUC therapy for the 24 weeks. After Week 24, participants continued NUC treatment during the follow-up unless the NUC discontinuation criteria were met.
- Combo 8: siRNA + PD-L1 LNA + NUC: Participants received siRNA, 200 mg, as a SC injection, Q4W up to Week 24 and PD-L1 LNA, 2 mg/kg, as a SC injection, QW during Weeks 25-36 in addition to their background NUC therapy for the 36 weeks. After Week 36, participants continued NUC treatment during the follow-up unless the NUC discontinuation criteria were met.
Arm/Group | NUC Control Arm | Combo 1: CpAM + TLR7 Agonist + NUC | Combo 2: siRNA (100 mg) + NUC | Combo 3: siRNA (200 mg) + NUC | Combo 4: siRNA + PEG-IFN + NUC | Combo 5: siRNA + CpAM + NUC | Combo 6: siRNA + TLR7 Agonist + NUC | Combo 7: siRNA + PD-L1 LNA + NUC | Combo 8: siRNA + PD-L1 LNA + NUC
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 12 | 7 | 10 | 9 | 5
percentage of participants
  Week 12 | 0 | 0 | 22.2 | 50 | 33.3 | 28.6 | 30 | 11.1 | 40
  Week 24: number analyzed (Participants) | 7 | 8 | 8 | 8 | 12 | 2 | 7 | 9 | 5
  Week 24 | 0 | 0 | 37.5 | 50 | 41.7 | 50 | 28.6 | 11.1 | 40
  Week 36: number analyzed (Participants) | 7 | 5 | 9 | 4 | 9 | 0 | 10 | 0 | 5
  Week 36 | 14.3 | 0 | 44.4 | 25 | 55.6 |  | 50 |  | 40
  Week 48: number analyzed (Participants) | 8 | 5 | 9 | 8 | 11 | 2 | 10 | 0 | 0
  Week 48 | 12.5 | 20 | 44.4 | 62.5 | 54.5 | 50 | 50 |  |
  FUW 12: number analyzed (Participants) | 6 | 8 | 7 | 8 | 11 | 3 | 9 | 9 | 5
  FUW 12 | 16.7 | 0 | 42.9 | 62.5 | 54.5 | 33.3 | 44.4 | 11.1 | 20
  FUW 24: number analyzed (Participants) | 7 | 8 | 8 | 8 | 11 | 3 | 9 | 9 | 5
  FUW 24 | 14.3 | 0 | 12.5 | 50 | 36.4 | 66.7 | 44.4 | 11.1 | 60
  FUW 36: number analyzed (Participants) | 8 | 8 | 8 | 8 | 11 | 0 | 9 | 6 | 3
  FUW 36 | 12.5 | 0 | 12.5 | 50 | 27.3 |  | 33.3 | 0 | 66.7
  FUW 48: number analyzed (Participants) | 7 | 8 | 9 | 8 | 11 | 0 | 9 | 5 | 0
  FUW 48 | 14.3 | 25 | 33.3 | 50 | 27.3 |  | 44.4 | 0 |

5. Secondary Outcome: Percentage of Participants With HBeAg Seroconversion in Baseline HBeAg-positive Participants
Description: HBeAg seroconversion was defined as a negative /non-reactive HBeAg level and a positive anti-HBe antibody. Percentages have been rounded off.
Time Frame: Weeks 12, 24, 36, and 48; FUW 12, 24, 36, and 48
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | NUC Control Arm | Combo 1: CpAM + TLR7 Agonist + NUC | Combo 2: siRNA (100 mg) + NUC | Combo 3: siRNA (200 mg) + NUC | Combo 4: siRNA + PEG-IFN + NUC | Combo 5: siRNA + CpAM + NUC | Combo 6: siRNA + TLR7 Agonist + NUC | Combo 7: siRNA + PD-L1 LNA + NUC | Combo 8: siRNA + PD-L1 LNA + NUC
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 12 | 7 | 10 | 9 | 5
percentage of participants
  Week 12 | 0 | 0 | 11.1 | 0 | 8.3 | 14.3 | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 7 | 8 | 8 | 8 | 12 | 2 | 7 | 9 | 5
  Week 24 | 0 | 0 | 0 | 12.5 | 8.3 | 0 | 0 | 0 | 0
  Week 36: number analyzed (Participants) | 7 | 5 | 9 | 4 | 9 | 0 | 10 | 0 | 5
  Week 36 | 0 | 0 | 11.1 | 0 | 11.1 |  | 10 |  | 0
  Week 48: number analyzed (Participants) | 8 | 5 | 9 | 8 | 11 | 2 | 10 | 0 | 0
  Week 48 | 0 | 0 | 11.1 | 12.5 | 18.2 | 0 | 10 |  |
  FUW 12: number analyzed (Participants) | 6 | 8 | 7 | 8 | 11 | 3 | 9 | 9 | 5
  FUW 12 | 16.7 | 0 | 14.3 | 12.5 | 18.2 | 0 | 11.1 | 0 | 0
  FUW 24: number analyzed (Participants) | 7 | 8 | 8 | 8 | 11 | 3 | 9 | 9 | 5
  FUW 24 | 14.3 | 0 | 0 | 25 | 9.1 | 33.3 | 11.1 | 0 | 0
  FUW 36: number analyzed (Participants) | 8 | 8 | 8 | 8 | 11 | 0 | 9 | 6 | 3
  FUW 36 | 12.5 | 0 | 0 | 25 | 9.1 |  | 11.1 | 0 | 0
  FUW 48: number analyzed (Participants) | 7 | 8 | 9 | 8 | 11 | 0 | 9 | 5 | 0
  FUW 48 | 14.3 | 0 | 11.1 | 37.5 | 9.1 |  | 33.3 | 0 |

6. Secondary Outcome: Number of Participants With Hepatitis B Virus Deoxyribonucleic Acid (HBV DNA) < Lower Limit of Quantification (LLOQ), <200 IU/mL, and <2,000 IU/mL
Description: Chronic HBV infection is characterized by high levels of circulating HBV DNA. Therefore, HBV levels are indicative of virological response. At screening participants were on NUC therapy and had circulating HBV DNA levels below the assay LLOQ or below 20 IU/mL for at least 6 months. The emergence of a virological breakthrough (HBV DNA >100 IU/mL or >1 log increase from nadir) while on NUC therapy, or the emergence of a virological relapse (>2,000 IU/mL) in participants taken off NME combination and NUC therapy during follow-up, was monitored through the quantification of HBV DNA in plasma.
Time Frame: FUW 12, 24, 36, and 48
Population: mITT population included participants who were randomized and received at least one dose of each drug for their assigned treatment regimen. Overall number analyzed included participants with data available for analysis. Number analyzed included participants with data available for analysis at that specified timepoint. Different participants may have contributed data for each timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | NUC Control Arm | Combo 1: CpAM + TLR7 Agonist + NUC | Combo 2: siRNA (100 mg) + NUC | Combo 3: siRNA (200 mg) + NUC | Combo 4: siRNA + PEG-IFN + NUC | Combo 5: siRNA + CpAM + NUC | Combo 6: siRNA + TLR7 Agonist + NUC | Combo 7: siRNA + PD-L1 LNA + NUC | Combo 8: siRNA + PD-L1 LNA + NUC
Number analyzed (Participants) | 35 | 35 | 30 | 30 | 30 | 9 | 34 | 33 | 30
Participants
  FUW 12: OFF NUC (< LLOQ): number analyzed (Participants) | 1 | 0 | 5 | 6 | 5 | 0 | 10 | 3 | 5
  FUW 12: OFF NUC (< LLOQ) | 0 |  | 3 | 4 | 4 |  | 7 | 2 | 4
  FUW 12: OFF NUC (≥ LLOQ - < 200 IU/mL): number analyzed (Participants) | 1 | 0 | 5 | 6 | 5 | 0 | 10 | 3 | 5
  FUW 12: OFF NUC (≥ LLOQ - < 200 IU/mL) | 1 |  | 1 | 1 | 0 |  | 2 | 1 | 1
  FUW 12: OFF NUC (≥ 200 - < 2000 IU/mL): number analyzed (Participants) | 1 | 0 | 5 | 6 | 5 | 0 | 10 | 3 | 5
  FUW 12: OFF NUC (≥ 200 - < 2000 IU/mL) | 0 |  | 1 | 1 | 1 |  | 1 | 0 | 0
  FUW 12: OFF NUC (≥ 2000 IU/mL): number analyzed (Participants) | 1 | 0 | 5 | 6 | 5 | 0 | 10 | 3 | 5
  FUW 12: OFF NUC (≥ 2000 IU/mL) | 0 |  | 0 | 0 | 0 |  | 0 | 0 | 0
  FUW 12: ON NUC (< LLOQ): number analyzed (Participants) | 28 | 32 | 19 | 23 | 21 | 8 | 20 | 30 | 25
  FUW 12: ON NUC (< LLOQ) | 28 | 32 | 19 | 23 | 21 | 8 | 20 | 30 | 24
  FUW 12: ON NUC (≥ LLOQ - < 200 IU/mL): number analyzed (Participants) | 28 | 32 | 19 | 23 | 21 | 8 | 20 | 30 | 25
  FUW 12: ON NUC (≥ LLOQ - < 200 IU/mL) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  FUW 12: ON NUC (≥ 200 - < 2000 IU/mL): number analyzed (Participants) | 28 | 32 | 19 | 23 | 21 | 8 | 20 | 30 | 25
  FUW 12: ON NUC (≥ 200 - < 2000 IU/mL) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  FUW 12: ON NUC (≥ 2000 IU/mL): number analyzed (Participants) | 28 | 32 | 19 | 23 | 21 | 8 | 20 | 30 | 25
  FUW 12: ON NUC (≥ 2000 IU/mL) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  FUW 24: OFF NUC (< LLOQ): number analyzed (Participants) | 2 | 0 | 4 | 5 | 7 | 0 | 12 | 8 | 9
  FUW 24: OFF NUC (< LLOQ) | 0 |  | 2 | 3 | 6 |  | 5 | 5 | 6
  FUW 24: OFF NUC (≥ LLOQ - < 200 IU/mL): number analyzed (Participants) | 2 | 0 | 4 | 5 | 7 | 0 | 12 | 8 | 9
  FUW 24: OFF NUC (≥ LLOQ - < 200 IU/mL) | 1 |  | 2 | 0 | 0 |  | 5 | 2 | 1
  FUW 24: OFF NUC (≥ 200 - < 2000 IU/mL): number analyzed (Participants) | 2 | 0 | 4 | 5 | 7 | 0 | 12 | 8 | 9
  FUW 24: OFF NUC (≥ 200 - < 2000 IU/mL) | 0 |  | 0 | 2 | 1 |  | 2 | 1 | 1
  FUW 24: OFF NUC (≥ 2000 IU/mL): number analyzed (Participants) | 2 | 0 | 4 | 5 | 7 | 0 | 12 | 8 | 9
  FUW 24: OFF NUC (≥ 2000 IU/mL) | 1 |  | 0 | 0 | 0 |  | 0 | 0 | 1
  FUW 24: ON NUC (< LLOQ): number analyzed (Participants) | 27 | 35 | 24 | 24 | 20 | 9 | 21 | 24 | 21
  FUW 24: ON NUC (< LLOQ) | 27 | 35 | 22 | 24 | 20 | 9 | 21 | 24 | 21
  FUW 24: ON NUC (≥ LLOQ - < 200 IU/mL): number analyzed (Participants) | 27 | 35 | 24 | 24 | 20 | 9 | 21 | 24 | 21
  FUW 24: ON NUC (≥ LLOQ - < 200 IU/mL) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  FUW 24: ON NUC (≥ 200 - < 2000 IU/mL): number analyzed (Participants) | 27 | 35 | 24 | 24 | 20 | 9 | 21 | 24 | 21
  FUW 24: ON NUC (≥ 200 - < 2000 IU/mL) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  FUW 24: ON NUC (≥ 2000 IU/mL): number analyzed (Participants) | 27 | 35 | 24 | 24 | 20 | 9 | 21 | 24 | 21
  FUW 24: ON NUC (≥ 2000 IU/mL) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  FUW 36: OFF NUC (< LLOQ): number analyzed (Participants) | 1 | 0 | 3 | 5 | 6 | 0 | 9 | 5 | 6
  FUW 36: OFF NUC (< LLOQ) | 0 |  | 1 | 3 | 6 |  | 1 | 5 | 3
  FUW 36: OFF NUC (≥ LLOQ - < 200 IU/mL): number analyzed (Participants) | 1 | 0 | 3 | 5 | 6 | 0 | 9 | 5 | 6
  FUW 36: OFF NUC (≥ LLOQ - < 200 IU/mL) | 0 |  | 1 | 0 | 0 |  | 3 | 0 | 2
  FUW 36: OFF NUC (≥ 200 - < 2000 IU/mL): number analyzed (Participants) | 1 | 0 | 3 | 5 | 6 | 0 | 9 | 5 | 6
  FUW 36: OFF NUC (≥ 200 - < 2000 IU/mL) | 1 |  | 0 | 2 | 0 |  | 5 | 0 | 0
  FUW 36: OFF NUC (≥ 2000 IU/mL): number analyzed (Participants) | 1 | 0 | 3 | 5 | 6 | 0 | 9 | 5 | 6
  FUW 36: OFF NUC (≥ 2000 IU/mL) | 0 |  | 1 | 0 | 0 |  | 0 | 0 | 1
  FUW 36: ON NUC (< LLOQ): number analyzed (Participants) | 29 | 31 | 25 | 25 | 21 | 1 | 24 | 17 | 13
  FUW 36: ON NUC (< LLOQ) | 29 | 31 | 24 | 25 | 21 | 1 | 22 | 16 | 13
  FUW 36: ON NUC (≥ LLOQ - < 200 IU/mL): number analyzed (Participants) | 29 | 31 | 25 | 25 | 21 | 1 | 24 | 17 | 13
  FUW 36: ON NUC (≥ LLOQ - < 200 IU/mL) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0
  FUW 36: ON NUC (≥ 200 - < 2000 IU/mL): number analyzed (Participants) | 29 | 31 | 25 | 25 | 21 | 1 | 24 | 17 | 13
  FUW 36: ON NUC (≥ 200 - < 2000 IU/mL) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  FUW 36: ON NUC (≥ 2000 IU/mL): number analyzed (Participants) | 29 | 31 | 25 | 25 | 21 | 1 | 24 | 17 | 13
  FUW 36: ON NUC (≥ 2000 IU/mL) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  FUW 48: OFF NUC (< LLOQ): number analyzed (Participants) | 0 | 0 | 2 | 7 | 6 | 0 | 9 | 5 | 4
  FUW 48: OFF NUC (< LLOQ) |  |  | 0 | 5 | 3 |  | 3 | 4 | 1
  FUW 48: OFF NUC (≥ LLOQ - < 200 IU/mL): number analyzed (Participants) | 0 | 0 | 2 | 7 | 6 | 0 | 9 | 5 | 4
  FUW 48: OFF NUC (≥ LLOQ - < 200 IU/mL) |  |  | 1 | 0 | 3 |  | 4 | 1 | 1
  FUW 48: OFF NUC (≥ 200 - < 2000 IU/mL): number analyzed (Participants) | 0 | 0 | 2 | 7 | 6 | 0 | 9 | 5 | 4
  FUW 48: OFF NUC (≥ 200 - < 2000 IU/mL) |  |  | 1 | 2 | 0 |  | 2 | 0 | 1
  FUW 48: OFF NUC (≥ 2000 IU/mL): number analyzed (Participants) | 0 | 0 | 2 | 7 | 6 | 0 | 9 | 5 | 4
  FUW 48: OFF NUC (≥ 2000 IU/mL) |  |  | 0 | 0 | 0 |  | 0 | 0 | 1
  FUW 48: ON NUC (< LLOQ): number analyzed (Participants) | 30 | 28 | 27 | 23 | 21 | 1 | 23 | 10 | 8
  FUW 48: ON NUC (< LLOQ) | 30 | 28 | 27 | 23 | 21 | 1 | 23 | 10 | 7
  FUW 48: ON NUC (≥ LLOQ - < 200 IU/mL): number analyzed (Participants) | 30 | 28 | 27 | 23 | 21 | 1 | 23 | 10 | 8
  FUW 48: ON NUC (≥ LLOQ - < 200 IU/mL) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  FUW 48: ON NUC (≥ 200 - < 2000 IU/mL): number analyzed (Participants) | 30 | 28 | 27 | 23 | 21 | 1 | 23 | 10 | 8
  FUW 48: ON NUC (≥ 200 - < 2000 IU/mL) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  FUW 48: ON NUC (≥ 2000 IU/mL): number analyzed (Participants) | 30 | 28 | 27 | 23 | 21 | 1 | 23 | 10 | 8
  FUW 48: ON NUC (≥ 2000 IU/mL) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline in HBsAg, Anti-HBs, HBeAg, HBV Ribonucleic Acid (RNA) and HBV DNA Levels Over Time
Description: The serological markers of HBV infection include viral antigens (HBsAg & HBeAg) and antibody (anti-HBs). Changes in serological markers and efficacy biomarkers (HBV RNA) from baseline are reported. Change from baseline for HBV DNA was assessed in 'ON NUC' participants.
Time Frame: HBsAg, Anti-HBs, HBeAg & HBV RNA: Combo 1 to 6 and NUC arm: Weeks 24, 36, 48, FUW 24 and FUW 48; Combo 7: Week 24, FUW 24 & FUW 48; Combo 8: Weeks 24, 36, FUW 24 & FUW 48; HBV DNA: FUW 24 and FUW 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | NUC Control Arm | Combo 1: CpAM + TLR7 Agonist + NUC | Combo 2: siRNA (100 mg) + NUC | Combo 3: siRNA (200 mg) + NUC | Combo 4: siRNA + PEG-IFN + NUC | Combo 5: siRNA + CpAM + NUC | Combo 6: siRNA + TLR7 Agonist + NUC | Combo 7: siRNA + PD-L1 LNA + NUC | Combo 8: siRNA + PD-L1 LNA + NUC
Number analyzed (Participants) | 35 | 36 | 30 | 30 | 30 | 9 | 34 | 33 | 30
log10 IU/mL
  HBsAg: Week 24: number analyzed (Participants) | 34 | 36 | 28 | 29 | 28 | 4 | 18 | 33 | 30
  HBsAg: Week 24 | -0.08 (0.16) | -0.11 (0.26) | -1.49 (0.56) | -1.78 (0.59) | -1.89 (1.05) | -1.38 (0.41) | -1.74 (0.62) | -2.12 (0.73) | -1.8 (0.49)
  HBsAg: Week 36: number analyzed (Participants) | 33 | 23 | 24 | 19 | 22 | 1 | 34 | 0 | 30
  HBsAg: Week 36 | -0.08 (0.13) | -0.13 (0.23) | -1.52 (0.67) | -1.93 (0.47) | -2.14 (1.27) | -1.51 (NA) — Since only 1 participant was analyzed, standard deviation (SD) could not be calculated. | -1.71 (0.69) |  | -2.08 (0.63)
  HBsAg: Week 48: number analyzed (Participants) | 34 | 20 | 29 | 30 | 28 | 4 | 34 | 0 | 0
  HBsAg: Week 48 | -0.2 (0.52) | -0.09 (0.12) | -1.58 (0.63) | -1.93 (0.6) | -2.22 (1.16) | -1.3 (0.45) | -2.18 (0.86) |  |
  HBsAg: FUW 24: number analyzed (Participants) | 29 | 35 | 28 | 30 | 27 | 9 | 31 | 32 | 30
  HBsAg: FUW 24 | -0.19 (0.35) | -0.18 (0.31) | -1.19 (0.76) | -1.71 (0.75) | -1.71 (1.24) | -1.5 (0.89) | -1.47 (0.81) | -1.3 (0.7) | -1.46 (0.74)
  HBsAg: FUW 48: number analyzed (Participants) | 30 | 28 | 29 | 30 | 27 | 1 | 32 | 15 | 12
  HBsAg: FUW 48 | -0.25 (0.43) | -0.25 (0.36) | -0.89 (0.76) | -1.2 (0.84) | -1.28 (1.12) | -2.02 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | -1.01 (0.8) | -0.91 (0.69) | -1.14 (0.83)
  Anti-HBs: Week 24: number analyzed (Participants) | 34 | 36 | 28 | 29 | 28 | 4 | 18 | 33 | 30
  Anti-HBs: Week 24 | -0.01 (0.04) | -0.01 (0.08) | 0.06 (0.32) | 0 (0) | 0.03 (0.2) | 0.06 (0.13) | -0.01 (0.04) | 0.01 (0.12) | -0.03 (0.1)
  Anti-HBs: Week 36: number analyzed (Participants) | 34 | 23 | 24 | 19 | 22 | 1 | 34 | 0 | 30
  Anti-HBs: Week 36 | -0.01 (0.02) | -0.02 (0.09) | 0.06 (0.34) | 0 (0) | 0.3 (0.69) | 0 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | -0.07 (0.27) |  | -0.03 (0.11)
  Anti-HBs: Week 48: number analyzed (Participants) | 34 | 20 | 29 | 30 | 28 | 4 | 34 | 0 | 0
  Anti-HBs: Week 48 | 0 (0.01) | -0.04 (0.11) | 0.06 (0.35) | 0 (0) | 0.55 (0.96) | 0.01 (0.02) | -0.05 (0.27) |  |
  Anti-HBs: FUW 24: number analyzed (Participants) | 29 | 35 | 28 | 30 | 27 | 9 | 31 | 32 | 25
  Anti-HBs: FUW 24 | -0.02 (0.08) | -0.01 (0.06) | 0.05 (0.31) | 0.01 (0.05) | 0.63 (1.04) | 0.09 (0.2) | -0.02 (0.41) | 0.01 (0.1) | -0.06 (0.2)
  Anti-HBs: FUW 48: number analyzed (Participants) | 30 | 28 | 29 | 30 | 27 | 1 | 32 | 9 | 9
  Anti-HBs: FUW 48 | 0.04 (0.33) | -0.01 (0.04) | 0.01 (0.28) | 0.02 (0.12) | 0.41 (0.93) | 0 (NA) — Since only 1 participant was analyzed, SD could not be calculated. | 0.04 (0.49) | 0.09 (0.26) | 0.02 (0.07)
  HBeAg: Week 24: number analyzed (Participants) | 7 | 8 | 8 | 8 | 12 | 2 | 7 | 9 | 5
  HBeAg: Week 24 | -0.08 (0.1) | -0.04 (0.13) | -0.39 (0.16) | -0.4 (0.21) | -0.37 (0.19) | -0.19 (0.32) | -0.53 (0.3) | -0.47 (0.32) | -0.46 (0.15)
  HBeAg: Week 36: number analyzed (Participants) | 7 | 5 | 9 | 4 | 9 | 0 | 10 | 0 | 5
  HBeAg: Week 36 | -0.08 (0.14) | -0.05 (0.04) | -0.45 (0.2) | -0.53 (0.15) | -0.43 (0.2) |  | -0.65 (0.44) |  | -0.46 (0.26)
  HBeAg: Week 48: number analyzed (Participants) | 8 | 5 | 9 | 8 | 11 | 2 | 10 | 0 | 0
  HBeAg: Week 48 | -0.06 (0.15) | -0.06 (0.06) | -0.48 (0.18) | -0.48 (0.2) | -0.44 (0.19) | -0.28 (0.42) | -0.69 (0.44) |  |
  HBeAg: FUW 24: number analyzed (Participants) | 7 | 8 | 8 | 8 | 11 | 3 | 9 | 9 | 5
  HBeAg: FUW 24 | -0.19 (0.15) | -0.09 (0.12) | -0.02 (1.37) | -0.42 (0.22) | -0.33 (0.19) | -0.68 (0.73) | -0.56 (0.33) | -0.4 (0.37) | -0.51 (0.31)
  HBeAg: FUW 48: number analyzed (Participants) | 7 | 8 | 9 | 8 | 11 | 0 | 9 | 5 | 0
  HBeAg: FUW 48 | -0.36 (0.31) | -0.22 (0.11) | -0.14 (1.06) | -0.38 (0.19) | -0.3 (0.16) |  | -0.5 (0.38) | -0.42 (0.47) |
  HBV RNA: Week 24: number analyzed (Participants) | 9 | 11 | 10 | 14 | 14 | 2 | 10 | 33 | 6
  HBV RNA: Week 24 | 0.09 (0.43) | -1.19 (1.19) | -0.7 (0.34) | -0.95 (0.6) | -1.43 (0.89) | -1.34 (0.65) | -0.92 (0.92) | -1.17 (1.26) | -0.81 (0.55)
  HBV RNA: Week 36: number analyzed (Participants) | 9 | 6 | 9 | 9 | 9 | 0 | 15 | 0 | 6
  HBV RNA: Week 36 | 0.05 (0.3) | -1.66 (1.4) | -0.74 (0.41) | -0.73 (0.57) | -1.67 (0.9) |  | -0.76 (0.76) |  | -0.76 (0.56)
  HBV RNA: Week 48: number analyzed (Participants) | 10 | 6 | 11 | 15 | 14 | 2 | 15 | 0 | 0
  HBV RNA: Week 48 | -0.04 (0.32) | -1.66 (1.4) | -0.8 (0.48) | -0.94 (0.6) | -1.43 (0.95) | -1.32 (0.68) | -0.9 (0.81) |  |
  HBV RNA: FUW 24: number analyzed (Participants) | 9 | 11 | 11 | 15 | 14 | 4 | 13 | 10 | 6
  HBV RNA: FUW 24 | -0.25 (0.28) | -0.13 (0.12) | -0.68 (0.49) | -0.87 (0.59) | -0.64 (0.82) | -1.04 (0.63) | -0.51 (0.63) | -0.82 (0.75) | -0.81 (0.55)
  HBV RNA: FUW 48: number analyzed (Participants) | 8 | 8 | 11 | 15 | 14 | 0 | 14 | 4 | 2
  HBV RNA: FUW 48 | -0.43 (0.6) | -0.11 (0.19) | -0.6 (0.48) | -0.78 (0.55) | -0.85 (0.75) |  | -0.37 (0.52) | -0.98 (0.8) | -0.49 (0.57)
  HBV DNA: FUW 24: number analyzed (Participants) | 27 | 35 | 24 | 24 | 20 | 9 | 21 | 24 | 21
  HBV DNA: FUW 24 | NA (NA) — Mean and SD were not estimable due to all of the samples being below LLOQ. | NA (NA) — Mean and SD were not estimable due to all of the samples being below LLOQ. | NA (NA) — Mean and SD were not estimable due to all of the samples being below LLOQ. | NA (NA) — Mean and SD were not estimable due to all of the samples being below LLOQ. | NA (NA) — Mean and SD were not estimable due to all of the samples being below LLOQ. | NA (NA) — Mean and SD were not estimable due to all of the samples being below LLOQ. | NA (NA) — Mean and SD were not estimable due to all of the samples being below LLOQ. | NA (NA) — Mean and SD were not estimable due to all of the samples being below LLOQ. | NA (NA) — Mean and SD were not estimable due to all of samples being below LLOQ.
  HBV DNA: FUW 48: number analyzed (Participants) | 30 | 28 | 2 | 7 | 6 | 1 | 9 | 10 | 8
  HBV DNA: FUW 48 | NA (NA) — Mean and SD were not estimable due to all of the samples being below LLOQ. | NA (NA) — Mean and SD were not estimable due to all of the samples being below LLOQ. | NA (NA) — Mean and SD were not estimable due to all of the samples being below LLOQ. | NA (NA) — Mean and SD were not estimable due to all of the samples being below LLOQ. | NA (NA) — Mean and SD were not estimable due to all of the samples being below LLOQ. | NA (NA) — Mean and SD were not estimable due to all of the samples being below LLOQ. | NA (NA) — Mean and SD were not estimable due to all of the samples being below LLOQ. | NA (NA) — Mean and SD were not estimable due to all of the samples being below LLOQ. | NA (NA) — Mean and SD were not estimable due to all of samples being below LLOQ.

8. Secondary Outcome: Combos 7 and 8: Area Under the Plasma Concentration-time Curve Over the Dosing Interval at Week 1 (AUC1-0-168h) of PD-L1 LNA
Description: The AUC was predicted and summarized by modelling & simulation via the population pharmacokinetics (PopPK) method based on pre and post dose samples. As per planned analysis data was collected and reported in a pooled manner for Combos 7 and 8.
Time Frame: Predose on Day 1 and up to 168 hours post dose (Week 1)
Population: PK population included participants who received at least one dose of the PD-L1 LNA and had at least one evaluable post-baseline PK sample.
Measure: Mean (Standard Deviation); unit: hours*nanomoles/liters (hr*nmol/L)
Groups:
- Combo 7 and 8: siRNA + PD-L1 LNA + NUC: Participants received siRNA, 200 mg, as a SC injection, Q4W up to Week 24 and PD-L1 LNA, 2 mg/kg, as a SC injection, QW during Weeks 13-24 (Combo 7)/ Weeks 25-36 (Combo 8) in addition to their background NUC therapy for 24 weeks (Combo 7)/ 36 weeks (Combo 8). After Week 24/36, participants continued NUC treatment during follow-up unless the NUC discontinuation criteria were met.
Arm/Group | Combo 7 and 8: siRNA + PD-L1 LNA + NUC
Number analyzed (Participants) | 63
hours*nanomoles/liters (hr*nmol/L) | 1047 (273)

9. Secondary Outcome: Combos 7 and 8: Maximum Plasma Concentration (Cmax) at Week 1 (Cmax1-0-168h) of PD-L1 LNA
Description: The Cmax was predicted and summarized by modelling & simulation via the PopPK method based on pre and post dose samples. As per planned analysis data was collected and reported in a pooled manner for Combos 7 and 8.
Time Frame: Predose on Day 1 and up to 168 hours post dose (Week 1)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: nanomoles/liters (nmol/L)
Groups:
- Combo 7 and 8: siRNA + PD-L1 LNA + NUC: Participants received siRNA, 200 mg, as a SC injection, Q4W up to Week 24 and PD-L1 LNA, 2 mg/kg, as a SC injection, QW during Weeks 13-24 (Combo 7)/ Weeks 25-36 (Combo 8) in addition to their background NUC therapy for 24 weeks (Combo 7)/ 36 weeks (Combo 8). After Week 24/36 participants continued NUC treatment during follow-up unless the NUC discontinuation criteria were met.
Arm/Group | Combo 7 and 8: siRNA + PD-L1 LNA + NUC
Number analyzed (Participants) | 63
nanomoles/liters (nmol/L) | 163 (60.8)

10. Secondary Outcome: Combos 7 and 8: AUC Over the Dosing Interval at Week 12 (AUC12-0-168h) of PD-L1 LNA
Description: The AUC was predicted and summarized by modelling & simulation via the PopPK method based on pre and post dose samples. As per planned analysis data was collected and reported in a pooled manner for Combos 7 and 8.
Time Frame: Predose on Day 1 of Week 12 up to 168 hours post dose (Week 12)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hr*nmol/L
Arm/Group | Combo 7 and 8: siRNA + PD-L1 LNA + NUC
Number analyzed (Participants) | 63
hr*nmol/L | 1143 (286)

11. Secondary Outcome: Combos 7 and 8: Cmax at Week 12 (Cmax12-0-168h) of PD-L1 LNA
Description: as for outcome 9
Time Frame: Predose on Day 1 of Week 12 up to 168 hours post dose (Week 12)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Combo 7 and 8: siRNA + PD-L1 LNA + NUC
Number analyzed (Participants) | 63
nmol/L | 165 (60.9)

12. Secondary Outcome: Combos 2, 3, 4, 6, 7 and 8: Area Under the Plasma Concentration Time Curve (AUC) Over Days 1-28 of siRNA
Description: The AUC was predicted and summarized by modelling & simulation via the PopPK method based on pre and post dose samples.
Time Frame: Predose on Day 1 and 1-3 and 4-6 hours post dose each day, up to Day 28
Population: PK population included participants who received at least one dose of the siRNA and had at least one evaluable post-baseline PK sample.
Measure: Mean (Standard Deviation); unit: hours*nanograms/millilitres (hr*ng/mL)
Arm/Group | Combo 2: siRNA (100 mg) + NUC | Combo 3: siRNA (200 mg) + NUC | Combo 4: siRNA + PEG-IFN + NUC | Combo 6: siRNA + TLR7 Agonist + NUC | Combo 7: siRNA + PD-L1 LNA + NUC | Combo 8: siRNA + PD-L1 LNA + NUC
Number analyzed (Participants) | 30 | 30 | 30 | 34 | 33 | 31
hours*nanograms/millilitres (hr*ng/mL) | 4670 (1112) | 11098 (2499) | 11073 (2272) | 9831 (2215) | 9780 (1942) | 9110 (1418)

13. Secondary Outcome: Combos 2, 3, 4, 6, 7 and 8: Cmax Over Days 1-28 of siRNA
Description: The Cmax was predicted and summarized by modelling & simulation via the PopPK method based on pre and post dose samples.
Time Frame: Predose on Day 1 and 1-3 and 4-6 hours post dose each day, up to Day 28
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: nanograms/millilitres (ng/mL)
Groups:
- Combo 6: siRNA + TLR7 Agonist + NUC: Participants received siRNA, 200 mg, as a SC injection, Q4W for 48 weeks and TLR7 agonist, 150 mg tablets, orally, QOD during Weeks 13-24 and Weeks 37-48 in addition to their background NUC therapy for 48 weeks. After Week 48, participants continued NUC treatment during follow-up unless the NUC discontinuation criteria were met.
Arm/Group | Combo 2: siRNA (100 mg) + NUC | Combo 3: siRNA (200 mg) + NUC | Combo 4: siRNA + PEG-IFN + NUC | Combo 6: siRNA + TLR7 Agonist + NUC | Combo 7: siRNA + PD-L1 LNA + NUC | Combo 8: siRNA + PD-L1 LNA + NUC
Number analyzed (Participants) | 30 | 30 | 30 | 34 | 33 | 31
nanograms/millilitres (ng/mL) | 190 (116) | 463 (203) | 450 (168) | 408 (168) | 373 (149) | 311 (97)

14. Secondary Outcome: Combos 2, 3, 4, 6, 7 and 8: Area Under the Plasma Concentration Time Curve During the Dosing Interval (AUC Tau) Over Days 29-56 of siRNA
Description: The AUC tau was predicted and summarized by modelling & simulation via the PopPK method based on pre and post dose samples. Simulations for the dosing interval between Day 29 and Day 56 was done using population PK modeling informed by sparse PK samples collected on Days 1, 85, 169, 253, and 337 at predose, 1-3 hours, and 4-6 hours post dose.
Time Frame: From Day 29 up to Day 56
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Combo 2: siRNA (100 mg) + NUC | Combo 3: siRNA (200 mg) + NUC | Combo 4: siRNA + PEG-IFN + NUC | Combo 6: siRNA + TLR7 Agonist + NUC | Combo 7: siRNA + PD-L1 LNA + NUC | Combo 8: siRNA + PD-L1 LNA + NUC
Number analyzed (Participants) | 30 | 30 | 30 | 34 | 33 | 31
hr*ng/mL | 5401 (1245) | 12591 (2659) | 12623 (2428) | 11207 (2371) | 11216 (2068) | 10513 (1511)

15. Secondary Outcome: Combos 2, 3, 4, 6, 7 and 8: Cmax Over Days 29-56 of siRNA
Description: The Cmax was predicted and summarized by modelling & simulation via the PopPK method based on pre and post dose samples. Simulations for the dosing interval between Day 29 and Day 56 was done using population PK modeling informed by sparse PK samples collected on Days 1, 85, 169, 253, and 337 at predose, 1-3 hours, and 4-6 hours post dose.
Time Frame: From Day 29 up to Day 56
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Combo 2: siRNA (100 mg) + NUC | Combo 3: siRNA (200 mg) + NUC | Combo 4: siRNA + PEG-IFN + NUC | Combo 6: siRNA + TLR7 Agonist + NUC | Combo 7: siRNA + PD-L1 LNA + NUC | Combo 8: siRNA + PD-L1 LNA + NUC
Number analyzed (Participants) | 30 | 30 | 30 | 34 | 33 | 31
ng/mL | 192 (116) | 468 (204) | 454 (169) | 411 (169) | 376 (150) | 315 (98)

16. Secondary Outcome: Combos 1 and 6: AUC of TLR7
Description: The AUC was predicted and summarized by modelling & simulation via the PopPK method based on pre and post dose samples.
Time Frame: Predose and 1-3 and 4-6 hours post-dose on Days 1, 3, 5 on Weeks 12 and 36
Population: PK population included participants who received at least one dose of the TLR7 and had at least one evaluable post-baseline PK sample.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Combo 1: CpAM + TLR7 Agonist + NUC | Combo 6: siRNA + TLR7 Agonist + NUC
Number analyzed (Participants) | 38 | 34
ng*hr/mL | 3139 (938.8) | 2813 (75.33)

17. Secondary Outcome: Combos 1 and 6: Cmax of TLR7
Description: The Cmax was predicted and summarized by modelling & simulation via the PopPK method based on pre and post dose samples.
Time Frame: Predose and 1-3 and 4-6 hours post-dose on Days 1, 3, 5 on Weeks 12 and 36
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Combo 1: CpAM + TLR7 Agonist + NUC | Combo 6: siRNA + TLR7 Agonist + NUC
Number analyzed (Participants) | 38 | 34
ng/mL | 1548 (419.7) | 1491 (334.8)

18. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product.
Time Frame: From Day 1 up to end of 48 weeks of follow up (up to approximately 1.8 years)
Population: Safety population included participants randomized to a treatment regimen who received at least one dose of any drug for their assigned treatment regimen, whether prematurely withdrawn from the study or not.
Measure: Count of Participants; unit: Participants
Arm/Group | NUC Control Arm | Combo 1: CpAM + TLR7 Agonist + NUC | Combo 2: siRNA (100 mg) + NUC | Combo 3: siRNA (200 mg) + NUC | Combo 4: siRNA + PEG-IFN + NUC | Combo 5: siRNA + CpAM + NUC | Combo 6: siRNA + TLR7 Agonist + NUC | Combo 7: siRNA + PD-L1 LNA + NUC | Combo 8: siRNA + PD-L1 LNA + NUC
Number analyzed (Participants) | 35 | 38 | 30 | 30 | 30 | 19 | 34 | 33 | 31
Participants | 27 | 34 | 30 | 29 | 30 | 18 | 33 | 26 | 27

19. Secondary Outcome: Combos 2, 3, 4, 5, 6, 7 and 8: Number of Participants With Anti-siRNA Antibodies
Description: Treatment-emergent anti drug antibody (ADA) was defined as participants who seroconverted or experienced a boost in preexisting ADA during the study. Participants were considered to be ADA positive if they were ADA negative or had missing data at baseline but develop an ADA response following study drug administration (treatment-induced ADA response), or if they were ADA positive at baseline and the titer of one or more post-baseline samples were greater than the titer of the baseline sample by a scientifically reasonable margin such as at least 4-fold (treatment-enhanced ADA response).
Time Frame: From Day 1 up to end of follow up (up to approximately 4 years)
Population: Immunogenicity population included participants who had at least one pre-dose (baseline) or at least one post-dose assessment will be included and analyzed according to the treatment they actually received or were allocated to receive.
Measure: Count of Participants; unit: Participants
Arm/Group | Combo 2: siRNA (100 mg) + NUC | Combo 3: siRNA (200 mg) + NUC | Combo 4: siRNA + PEG-IFN + NUC | Combo 5: siRNA + CpAM + NUC | Combo 6: siRNA + TLR7 Agonist + NUC | Combo 7: siRNA + PD-L1 LNA + NUC | Combo 8: siRNA + PD-L1 LNA + NUC
Number analyzed (Participants) | 30 | 30 | 30 | 19 | 34 | 33 | 31
Participants | 3 | 2 | 12 | 1 | 3 | 10 | 14

20. Secondary Outcome: Combos 7 and 8: Number of Participants With Anti-PD-L1 Antibodies
Description: Treatment-emergent ADA was defined as participants who seroconverted or experienced a boost in preexisting ADA during the study. Participants were considered to be ADA positive if they were ADA negative or had missing data at baseline but develop an ADA response following study drug administration (treatment-induced ADA response), or if they were ADA positive at baseline and the titer of one or more post-baseline samples were greater than the titer of the baseline sample by a scientifically reasonable margin such as at least 4-fold (treatment-enhanced ADA response).
Time Frame: From Day 1 for Combo 7 and 8 up to end of follow up (Up to approximately 2 years)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Combo 7: siRNA + PD-L1 LNA + NUC | Combo 8: siRNA + PD-L1 LNA + NUC
Number analyzed (Participants) | 33 | 31
Participants | 16 | 15

ADVERSE EVENTS:
Time Frame: From Day 1 up to end of 48 week follow up (up to approximately 1.8 years)
Description: Safety population included participants randomized to a treatment regimen who received at least one dose of any drug for their assigned treatment regimen, whether prematurely withdrawn from the study or not.
Arm/Group | Combo 1: CpAM + TLR7 Agonist + NUC | Combo 2: siRNA (100 mg) + NUC | Combo 3: siRNA (200 mg) + NUC | Combo 4: siRNA + PEG-IFN + NUC | Combo 5: siRNA + CpAM + NUC | Combo 6: siRNA + TLR7 Agonist + NUC | Combo 7: siRNA + PD-L1 LNA + NUC | Combo 8: siRNA + PD-L1 LNA + NUC | NUC Control Arm
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/30 | 0/30 | 0/30 | 0/19 | 0/34 | 0/33 | 0/31 | 0/35
Serious Adverse Events (participants affected / at risk) | 3/38 | 3/30 | 4/30 | 2/30 | 0/19 | 2/34 | 0/33 | 0/31 | 1/35
Other Adverse Events (participants affected / at risk) | 33/38 | 27/30 | 29/30 | 29/30 | 18/19 | 33/34 | 23/33 | 25/31 | 25/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combo 1: CpAM + TLR7 Agonist + NUC (N=38) | Combo 2: siRNA (100 mg) + NUC (N=30) | Combo 3: siRNA (200 mg) + NUC (N=30) | Combo 4: siRNA + PEG-IFN + NUC (N=30) | Combo 5: siRNA + CpAM + NUC (N=19) | Combo 6: siRNA + TLR7 Agonist + NUC (N=34) | Combo 7: siRNA + PD-L1 LNA + NUC (N=33) | Combo 8: siRNA + PD-L1 LNA + NUC (N=31) | NUC Control Arm (N=35)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fascioliasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic reaction (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combo 1: CpAM + TLR7 Agonist + NUC (N=38) | Combo 2: siRNA (100 mg) + NUC (N=30) | Combo 3: siRNA (200 mg) + NUC (N=30) | Combo 4: siRNA + PEG-IFN + NUC (N=30) | Combo 5: siRNA + CpAM + NUC (N=19) | Combo 6: siRNA + TLR7 Agonist + NUC (N=34) | Combo 7: siRNA + PD-L1 LNA + NUC (N=33) | Combo 8: siRNA + PD-L1 LNA + NUC (N=31) | NUC Control Arm (N=35)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Monocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 0 (0) | 5 (5) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 2 (3) | 3 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 1 (1) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (2) | 3 (4) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 4 (5) | 4 (4) | 1 (2) | 1 (1) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (2) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (3) | 2 (8) | 1 (1) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Fatigue (General disorders) | 5 (5) | 1 (1) | 2 (2) | 7 (12) | 1 (1) | 3 (3) | 3 (8) | 3 (3) | 0 (0)
Influenza like illness (General disorders) | 14 (62) | 0 (0) | 0 (0) | 8 (12) | 1 (1) | 16 (38) | 0 (0) | 4 (6) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 2 (2) | 9 (16) | 15 (39) | 3 (4) | 7 (10) | 5 (9) | 7 (37) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 6 (9) | 0 (0) | 3 (3) | 7 (7) | 4 (4) | 7 (10) | 1 (1) | 2 (2) | 1 (1)
Sensation of foreign body (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatic mass (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 7 (8) | 3 (3) | 6 (6) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 4 (4)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 6 (6) | 10 (10) | 16 (17) | 17 (17) | 3 (3) | 17 (18) | 3 (3) | 4 (4) | 8 (8)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis B reactivation (Infections and infestations) | 0 (0) | 6 (6) | 1 (1) | 2 (2) | 0 (0) | 10 (10) | 4 (4) | 7 (7) | 3 (3)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (5) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 14 (24) | 11 (16) | 13 (16) | 5 (6) | 4 (6) | 1 (1) | 2 (4) | 4 (4)
Accidental overdose (Injury, poisoning and procedural complications) | 8 (10) | 5 (5) | 6 (6) | 0 (0) | 1 (1) | 4 (6) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Product dose omission issue (Injury, poisoning and procedural complications) | 2 (3) | 13 (14) | 14 (14) | 19 (23) | 2 (7) | 15 (33) | 0 (0) | 0 (0) | 13 (13)
Alanine aminotransferase increased (Investigations) | 4 (5) | 13 (22) | 13 (21) | 25 (39) | 10 (16) | 15 (25) | 6 (6) | 6 (8) | 3 (3)
Amylase increased (Investigations) | 0 (0) | 5 (6) | 5 (5) | 6 (14) | 1 (1) | 5 (6) | 3 (3) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 6 (11) | 10 (17) | 21 (32) | 7 (7) | 11 (21) | 4 (4) | 2 (3) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (5) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 3 (8) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Cystatin C increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram PR shortened (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 7 (9) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Glutamate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 5 (12) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 3 (4) | 3 (5) | 2 (4) | 3 (5) | 2 (4) | 4 (4) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (4) | 1 (2) | 1 (3) | 12 (24) | 0 (0) | 6 (11) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 17 (26) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 8 (12) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroxine free decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 4 (4) | 1 (2) | 1 (4) | 8 (14) | 0 (0) | 5 (11) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 6 (10) | 7 (15) | 1 (1) | 0 (0) | 4 (11) | 0 (0) | 1 (1) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (4) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 6 (9) | 6 (9) | 3 (5) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 3 (4) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 2 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 3 (4) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (4) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 5 (12) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (24) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (6) | 2 (3) | 3 (4) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Prostatic calcification (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 5 (5) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT04225715/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT04225715/SAP_001.pdf